CLINICAL TRIAL: NCT00565994
Title: A Study of Cytokine and Inflammatory Markers in Patients With Chronic Renal Failure According to Their Method of Vascular Access
Brief Title: A Study of Cytokine and Inflammatory Markers in Patients With Chronic Renal Failure
Status: Completed | Type: Observational
Sponsor: University of Oklahoma (Other)
Responsible Party: William Jennings, MD, University of Oklahoma-Tulsa, Dept. of Surgery
Other Study IDs: OUHSC IRB #13137
Record Dates: First submitted 2007-11-29; First posted 2007-11-30 (Estimated); Last update posted 2010-09-28 (Estimated); Status verified 2010-09

CONDITIONS: Chronic Renal Failure
Keywords: hemodialysis; Vascular access; arteriovenous fistula; indwelling percutaneous catheters; arteriovenous grafts
MeSH Terms: conditions — Kidney Failure, Chronic; Arteriovenous Fistula | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Hemodialysis patients: Male and female patients undergoing hemodialysis therapy as outpatients
  Interventions: Procedure: Blood Draw
- Control: Male and female healthy volunteers
  Interventions: Procedure: Blood Draw
- Pre-dialysis patients: Male and female patients with Stage 3, 4, or 5 chronic kidney disease, but not yet on dialysis
  Interventions: Procedure: Blood Draw

INTERVENTIONS:
Procedure: Blood Draw — For patients undergoing routine hemodialysis for chronic renal failure, 5-10 ml of blood will be removed from the dialysis tubing during vascular access. All other subjects will have 5-10 ml of blood drawn by routine venipuncture.

SUMMARY:
We hope to study components within the blood that may predict success, failure or other associated complications in relation to the type of vascular access being used.

DETAILED DESCRIPTION:
Renal failure affects more than 350,000 patients in the United States. All patients undergoing dialysis must have access to the vascular system (blood stream) for hemodialysis treatment. Methods of access include a catheter, or tube, that goes through the skin and into a large vein, a surgically created connection of a vein to an artery called an AV fistula, or a surgically created connection of a vein to artery using a graft or plastic tube. Previous research has shown considerable differences in the function and success in these types of vascular access for dialysis. Research investigators try to explain these differences and find the causes and explanations for the variations seen in vascular access.

Forty patients undergoing dialysis treatment will be evaluated by analyzing serum specimens obtained during outpatient hemodialysis access. Serum will also be collected from ten pre-dialysis patients and ten normal volunteers for comparison. Pre-dialysis patients are those who have Stage 3, 4, or 5 chronic kidney disease but are not yet on dialysis and have never had any type of created vascular access. Normal subjects will have no kidney disease, autoimmune disorders, recent (<6 months) chemotherapy treatment or corticosteroid use, or other chronic condition determined by the investigator to interfere with cytokine and inflammatory markers. The serum specimens will be analyzed for cytokine/inflammatory markers and correlated with clinical access type and other medical data and demographic information.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients of Dr. William Jennings and Dr. Pranay Kathuria undergoing dialysis therapy as outpatients
* Male and female patients of Dr. Pranay Kathuria who have been diagnosed with Stage 3, 4, or 5 chronic kidney disease, but who are not yet on dialysis.
* Healthy volunteers with no kidney disease, autoimmune disorders, recent (<6 months) chemotherapy treatment or corticosteroid use, or other chronic condition determined by the investigator to interfere with cytokine and inflammatory markers.
* 18 to 90 years of age

Exclusion Criteria:

* under 18 years of age
* over 90 years of age
* prisoners
* institutionalized patients
* pregnant individuals
* patients with mental illness who are not able to give informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female patients of Dr. William Jennings and Dr. Pranay Kathuria undergoing dialysis therapy as outpatients. Dialysis and pre-dialysis patients will be recruited from Dr. Pranay Kathuria's practice. Normal volunteers will be recruited from family members of the pre-dialysis patients, Internal Medicine patients already scheduled to have blood drawn for other reasons, or from faculty/staff/student volunteers who are not otherwise involved with the study and are not in a subordinate role to any of the study investigators.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2008-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William C Jennings, MD, Principal Investigator — University of Oklahoma-Tulsa
Locations (1):
- University of Oklahoma-Tulsa, Tulsa, Oklahoma, United States